CLINICAL TRIAL: NCT01670123
Title: Development of a Personalized Real-time Intervention for Bipolar Disorder
Acronym: PRISM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Colin Depp, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MH091260
Record Dates: First submitted 2012-08-17; First posted 2012-08-21 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Bipolar Disorder
Keywords: Mobile phone; electronic intervention; behavioral intervention; telehealth; bipolar disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mobile Phone Condition (Experimental): This arm will involve daily self-monitoring with an electronic mobile device with responses to survey questions about mood status. Mood status reports are linked with personalized coping strategies.
  Interventions: Behavioral: Personalized Real-Time Intervention for Stabilizing Mood
- Paper-and-pencil condition (Placebo Comparator): This arm will complete a paper-and-pencil mood chart on a daily basis
  Interventions: Behavioral: Personalized Real-Time Intervention for Stabilizing Mood

INTERVENTIONS:
Behavioral: Personalized Real-Time Intervention for Stabilizing Mood — Interactive mobile web-based behavioral intervention targeting symptoms of bipolar disorder

SUMMARY:
This three-year intervention development proposal is submitted to the NIMH DATR Mood Disorders/Sleep Disorders Program A2-AID and is led by a New Investigator. The goal of this study is to further develop and then evaluate the clinical utility of a new personalized smart-phone intervention to enhance illness self-management in people with bipolar disorder. Bipolar disorder is a heterogeneous fluctuating condition and a leading source of disability. Consistent with NIMH Strategic Aim 3.2, self-monitoring tools are vital to clinical management and evidence-based psychosocial interventions for bipolar disorder. Practice guidelines state that all patients should receive education in self-monitoring and identifying adaptive responses to early warning signs and symptoms. Advances in technology have enabled electronic monitoring of patient-reported outcomes using mobile devices - an assessment strategy called Ecological Momentary Assessment (EMA). Using freely available software, we have developed a preliminary version of a novel smart-phone intervention that integrates EMA with brief psychosocial intervention designed for people with bipolar disorder. Mobile real-time interventions have been successfully applied in other chronic illnesses and have theoretical advantages over clinic-based interventions in motivating and cuing health-protective behavior. Our new intervention is called Personalized Real-Time Intervention for Stabilizing Mood (PRISM), and it delivers tailored intervention content naturalistically at the moment that symptoms occur. We recently conducted a small proof-of-concept study of PRISM in outpatient adults with bipolar disorder that suggests the intervention is feasible, presents no technological or operational barriers, yields data that corresponds with clinical ratings, and is perceived as useful by participants. Building from our preliminary work, we propose to further develop the intervention based on participant feedback and theoretically-driven enhancements. We will then conduct a randomized trial to assess the clinical utility of this new intervention over 12 weeks. Specifically, we will randomize a sample of 90 adults aged 18 and older with Bipolar Disorder I or II to one of two experimental conditions. Participants in both conditions will participate in two in-person sessions adapted from an evidence-based psychosocial intervention for bipolar disorder, aimed at identifying early warning signs and adaptive responses to symptom fluctuations. The Control condition will participate in the in-person sessions, and the PRISM condition will also utilize the smart phone device for 12 weeks. In this pilot trial, we will compare outcomes between the two conditions on standard clinical ratings of depressive and manic symptoms, along with psychosocial functioning. We will assess predictors of compliance and changes in outcomes in the PRISM condition to inform a larger effectiveness trial. We will use exploratory analyses to further refine the intervention, including capitalizing on the rich repeated measures obtained by the device. This study will provide a strong basis for a larger effectiveness trial, along with a potentially useful tool to enhance self-management in bipolar disorder. PUBLIC HEALTH RELEVANCE: Bipolar disorder is a leading cause of disability, and many people do not have access to evidence-based psychosocial interventions. Mobile devices may prove more effective than clinic-based interventions, because they deliver self-management strategies at the moment that symptoms occur. To lead to a larger effectiveness study, we propose to further develop our novel intervention uses mobile technology to monitor and intervene with symptoms in real-time, and then conduct a 12-week randomized trial in 90 patients to evaluate the acceptability and short-term efficacy of our smart-phone based intervention for bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of bipolar disorder
* Currently an outpatient

Exclusion Criteria:

* Psychiatric hospitalization in the past month
* Substance abuse diagnosis in the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale | 3 month
  Depression severity measure

SECONDARY OUTCOMES:
Young Mania Rating Scale | 3 Month
  Mania symptom severity

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, La Jolla, California, United States

REFERENCES:
- [Derived] Depp CA, Kim DH, de Dios LV, Wang V, Ceglowski J. A Pilot Study of Mood Ratings Captured by Mobile Phone Versus Paper-and-Pencil Mood Charts in Bipolar Disorder. J Dual Diagn. 2012 Jan 1;8(4):326-332. doi: 10.1080/15504263.2012.723318. PMID 23646035